CLINICAL TRIAL: NCT02242162
Title: Establishment of a Non-invasive and Indirect Measure of Volitional Pimax
Acronym: PI MAX STIM
Status: Completed | Type: Observational
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Sponsor
Other Study IDs: 2009-A00630-57
Record Dates: First submitted 2014-09-15; First posted 2014-09-16 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-03

CONDITIONS: Neuromuscular Diseases; Respiratory Failure
Keywords: phrenic nerves magnetic stimulations
MeSH Terms: conditions — Neuromuscular Diseases; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- neuromuscular diseases
  Interventions: Procedure: phrenic nerves magnetic stimulations

INTERVENTIONS:
Procedure: phrenic nerves magnetic stimulations

SUMMARY:
Respiratory failure is the main death cause in muscular diseases. Non-invasive and volitional measures of inspiratory muscles strength include the nasal pressure with an occluded nostril and the maximal inspiratory pressure (PImax).Unfortunately, volitional maneuvers depend of patient effort. The mean of this reseach is to validate a non-invasive and non-volitional technique to evaluate diaphragm strength at muscular diseases patients.The methdology consist to compar PImax measure to nerves magnetical stimulation maneuvers measure.

ELIGIBILITY:
Inclusion Criteria:

* Neuromuscular disease
* Pimax evaluation indication

Exclusion Criteria:

* pregnant women
* usual contre-indications for nuclear magnetic resonance

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: neuromuscular diseases
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2009-05; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
magnetic stimulation pressure measure( Pstim) | 10 minutes
  phrenic nerves magnetic stimulations

CONTACTS AND LOCATIONS:
Overall Officials: frederic Lofaso, Pr, Principal Investigator — Hopital R Poincaré
Locations (1):
- Hopital R Poincaré, Garches, France